CLINICAL TRIAL: NCT04600765
Title: Clinical Blood Profile Assays as Biomarkers to Directly Assess Potential Health Effects Resulting From the Controlled Elimination of Suspected Dietary and Environmental Chemical Toxins
Brief Title: hsCRP Clinical Inflammation Marker for Human Bisphenol A Food Contamination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Research on Environmental Chemicals in Humans (Other)
Responsible Party: Principal Investigator, William Lewis Perdue III, Chairman, Center for Research on Environmental Chemicals in Humans
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UCSF-IRB-IRB-15-17703
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diet Before (Active Comparator): Typical diet contaminated with Bisphenol A. Patient assigned to this arm will consume a typical American diet as defined by USDA.
  Interventions: Diagnostic Test: hsCRP serum measurement of inflammation
- Diet After (Active Comparator): Bisphenol A reduced. Patient assigned to this arm will consume a diet analogous to atypical American diet as defined by USDA, but with known Bisphenol A sources reduced or eliminated.
  Interventions: Diagnostic Test: hsCRP serum measurement of inflammation

INTERVENTIONS:
Diagnostic Test: hsCRP serum measurement of inflammation — hsCRP inflammation change as result of non-contaminated diet

SUMMARY:
Dietary intervention studies thus far have failed to be replicable or causal.This is particularly relevant regarding plastic-derived chemicals (PDCs),This first-of-a-kind dietary intervention study explores a potential causal relationship between human serum levels of BPA and High-Sensitivity C-Reactive Protein (hsCRP)

DETAILED DESCRIPTION:
Dietary intervention studies thus far have failed to be replicable or causal. The results, therefore, have failed to provide clinicians and the general public with consistent and useful information on which to base reliable food-related health decisions. This is particularly relevant regarding plastic-derived chemicals (PDCs), such as Bisphenol A, now that the federal CLARITY-BPA program has failed to achieve scientific consensus. Investigators propose a novel human dietary protocol that is both replicable and causal, based upon BPA's demonstrated inflammatory effects in humans. This first-of-a-kind dietary intervention study explores a potential causal relationship between human serum levels of BPA and High-Sensitivity C-Reactive Protein (hsCRP), a proven clinical indicator of inflammation. Investigators used the equivalent of a USDA-defined "typical diet" followed by a PDC-reduced diet to compare blood levels of hsCRP. This proof-of-concept investigation is the first to use an easily accessible, medically-accepted clinical laboratory test to directly measure human health effects of PDC reduction. Unexpected new complications discovered during the investigation indicate that these results may yet be inconclusive for direct causal relationship. However, the novel lessons and techniques developed as a result of those discoveries offer further specific and improved methods and best practices that can enable future dietary interventions to produce replicable, causal results.

ELIGIBILITY:
INCLUSION CRITERIA

* Overall good health
* hsCRP below 10
* Standard health review blood panel normal
* BMI less than 25
* % body fat less than 23%
* Resident of North San Francisco Bay area
* Willing to eat 100% of all foods and beverages provided.
* No food allergies
* Not taking prescription medications or supplements including daily aspirin.
* Written unformed consent
* Any one not compliant with inclusion criteria.

EXCLUSION CRITERIA

* Subject in poor health
* hsCRP above 10
* Standard health review blood panel beyond minimum or maximum limits for any measurement.
* Taking taking prescription medications or supplements including daily aspirin.
* Any evidence of inflammation-linked disease or syndrome including cardiovascular, metabolic syndrome, Type 2 Diabetes, insulin resistance, obesity, auto-immune disease, depression, or other neurological or behavioral disorders.

Ages: 60 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 1 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
hsCRP Serum concentration vs serum Bisphenol A concentration | 6 days
  Will decreasing Bisphenol A concentration in subject diet alter inflammatinn measure

CONTACTS AND LOCATIONS:
Overall Officials: WILLIAM L PERDUE, Principal Investigator — Center for Research on Environmental Chemicals in Humans; Victor I Reus, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Center for Research on Environmental Chemicals in Humans, Sonoma, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Because this is an n-of-1, proof of concept study, all data will be share upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- See also: Site for posting study-related information, preliminary findings, and supplemental information. — https://stealthsyndromestudy.com
- See also: Site for the Center for Research on Environmental Chemicals in Humans -- the 501(c)(3) non-profit supporting this study. — https://crechcenter.org